CLINICAL TRIAL: NCT06576960
Title: Caries Inhibitory Effect of Nano Silver Varnish Versus Tri Calcium Phosphate Varnish Among Children With Visual Impairment
Brief Title: Caries Inhibitory Effect of Nano Silver and Tri Calcium Phosphate Varnishes Among Visually Impaired Children
Acronym: Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadeer Mohammed Abd El wahab (Other)
Collaborators: Tanta University (Other)
Responsible Party: Sponsor-Investigator, Hadeer Mohammed Abd El wahab, El Mahalla Elkobra, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OH12-12
Record Dates: First submitted 2024-08-26; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- nano silver varnish (Experimental): new fluoride varnish
  Interventions: Drug: Nano silver fluoride varnish and tri calcium phosphate varnish
- tri calcium phosphate varnish (Experimental): fluoride varnish contain calcium phosphate
  Interventions: Drug: Nano silver fluoride varnish and tri calcium phosphate varnish
- health education (No Intervention)

INTERVENTIONS:
Drug: Nano silver fluoride varnish and tri calcium phosphate varnish — Fluoride varnishes
  Other Names: health education
  Arms: nano silver varnish; tri calcium phosphate varnish

SUMMARY:
Assessment of pH,streptococcus mutants count, lactobacillus count and immunoglobulin A among visually impaired children after nano silver varnish application it tri calcium phosphate phosphate varnish application

DETAILED DESCRIPTION:
Sixty children will be randomly divided into three equal treatment groups, composed of 20 children each, according to the type of material used as follows:

* Group I: children will receive oral health education and nano silver fluoride varnish.
* Group II: children will receive oral health education and tri calcium phosphate varnish.
* Group III: children will receive oral health education

for all children ,Assessment of pH, streptococcus mutants count, lactobacillus count and immunoglobulin A will be assessed at baseline, one day , 3 months and 6 months after application

ELIGIBILITY:
Inclusion Criteria:

Visually impaired children

Exclusion Criteria:

* uncooperative children or children not willing to participate in the study.
* Children with systemic diseases
* Children with bronchial asthma.
* Children who were on antibiotic or medications that might affect oral flora or salivary flow taken within the previous 3 months
* History of fluoride treatment in the past 3-4 weeks.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-04-13 (Actual)

PRIMARY OUTCOMES:
Salivary PH | 6 months
  Salivary power of hydrogen at baseline, one month, 3months and six months after intervention
Salivary streptococcus mutants count | 6months
  Count of bacteria at baseline, one day, 3months and six months after intervention
Lactobacillus count | 6 months
  Count of bacteria at baseline, one day, 3months and six months after intervention
Immunoglobulin A | 6months
  Level of immunoglobulin A at saliva at baseline, one day, 3months and 6 months after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Amin, PhD, Study Director — Faculty of dentistry . Tanta university
Locations (1):
- Faculty of dentistry, Tanta, Tanta City, Egypt

IPD SHARING:
Plan to Share IPD: No